CLINICAL TRIAL: NCT03070002
Title: A Phase II, Open Label Study to Evaluate Denosumab in Patients With ER and/or PR-Positive, HER2-Negative Metastatic Breast Cancer (MBC) With Bone Metastases and Detectable Circulating Tumor Cells (CTCs)
Brief Title: Denosumab in Treating Patients With ER and/or PR Positive, HER2 Negative Metastatic Breast Cancer With Bone Metastases and Detectable Circulating Tumor Cells
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Northwestern University (Other)
Collaborators: Amgen (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16B09; STU00203216 (CTRP (Clinical Trial Reporting Program)); NU 16B09 (Other: Northwestern University); P30CA060553 (NIH); NCI-2017-00015 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Breast Carcinoma Metastatic in the Bone; Circulating Tumor Cell Count; Estrogen Receptor Positive; HER2/Neu Negative; Progesterone Receptor Positive; Stage IV Breast Cancer
MeSH Terms: conditions — Neoplastic Cells, Circulating; Breast Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (denosumab) (Experimental): Patients receive denosumab SC on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression, unexpected toxicity, or patient withdrawal or death.
  Interventions: Biological: Denosumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Denosumab — Given SC
  Other Names: AMG 162; AMG-162; Prolia; Xgeva
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
The purpose of this study is to look at the amount of cancer cells in the blood of participants who are being treated with denosumab. The other purpose is to look at how long it takes for cancer to get worse when participants are being treated with denosumab. Circulating tumor cells (CTCs) in the blood of patients with metastatic breast cancer (MBC) have been associated with shorter survival than when CTCs are absent, especially in patients whose cancer has spread to their bones. In this study, we want it see if denosumab (the study drug) will decrease the number of CTCs measured in patients with MBC and cancer that has spread to their bones. We also plan to get blood from participants to study other research markers of interest.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the effect of denosumab in Her2/neu negative ER+ and/or PR+ metastatic breast cancer patients who are in partial response (PR) or stable disease (SD) after starting systemic therapy with bone metastases and >= 5 circulating tumor cells (CTCs) by measuring the fraction of patients with reduction in CTCs after 3 cycles of denosumab.

SECONDARY OBJECTIVES:

I. To assess the effect of denosumab on CTCs enumeration considered as a continuous variable (percent change from baseline) in this population.

II. To evaluate median progression-free survival (m-PFS).

TERTIARY OBJECTIVES:

I. CTC enumeration after enrichment. II. To assess the effect on CTC profiling and characterization of stem cell phenotype (CTC-EMT).

III. To evaluate the type of progressive disease (new site versus [vs.] progression of lesions in previous sites).

IV. To analyze the expression of RANKL.

OUTLINE:

Patients receive denosumab subcutaneously (SC) on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression, unexpected toxicity, or patient withdrawal or death.

After completion of study treatment, patients are followed up every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed ER and/or PR positive, HER-2/neu negative metastatic breast cancer; they can be enrolled in any line of therapy without investigational agents and should have stable disease or a partial response (which can be determined clinically) on current systemic treatment; patients must also have pathologic OR radiographic evidence of bone metastases and >= 5 CTCs; (Note: the pathology report that is used by the physician to determine diagnosis, will be used to determine patient eligibility; ER and PR status should be available at the time of registration)
* Patients may have either measurable or non-measurable within 30 of days of registration; (lesions treated with radiation therapy must not be used as a target lesion); (Note: per Response Evaluation Criteria in Solid Tumors [RECIST] criteria version [v.] 1.1, measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension; non-measurable disease is defined as all other lesions, including small lesions [longest diameter < 10 mm or pathological lymph nodes with P10 to < 15 mm short axis] as well as truly non-measurable lesions; lesions considered truly nonmeasurable include: leptomeningeal disease, ascites, pleural or pericardial effusion, and inflammatory breast disease, lymphangitic involvement of skin or lung, abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques)
* Patients may be enrolled in any line of standard treatment (without investigational agents); the start date of current treatment should be at least two 2 weeks or more prior to registration; (Note: patients will continue to receive the planned active treatment with chemotherapy or endocrine therapy [standard of care] and initiate denosumab at the recommended dose for this protocol)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Leukocytes >= 3,000/mcL (without growth factor)
* Platelets >= 100,000/mcL (with or without transfusion)
* Hemoglobin >= 8 (with or without transfusion)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (serum glutamic-oxaloacetic transaminase [SGOT] and serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times institutional upper limit of normal (for patients with liver metastasis up to =< 5 times of upper limit of normal [ULN] is allowed)
* Bilirubin =< 1.5 ULN (for patients with liver metastasis up to =< 5 times of ULN is allowed)
* Serum creatinine =< 1.5 ULN
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (creatinine clearance should be calculated per institutional standard)
* Patients must have a serum calcium of >= 2.0 mmol/L (8.0 mg/dL) or albumin-adjusted serum calcium =< 2.9 mmol/L (11.5 mg/dL) within 30 days of registration; (Note: if patients are undergoing treatment for hypocalcemia and the serum calcium value at screening is > 8.0 mg/dl, then the patient will be eligible for this study)
* Females of child-bearing potential (FOCBP) and males with his or her partner must agree to use two acceptable methods of effective contraception, at study entry, for the duration of study participation, and for 5 months following completion of therapy; subjects who are surgically sterile (e.g., history of bilateral tubal ligation, hysterectomy) or whose sexual partner is sterile (e.g., history of vasectomy) are not required to use additional contraceptive measures; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; likewise, if a male patient impregnates his female partner, he should inform the treating physician immediately; NOTE: a FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative serum OR urine pregnancy test =< 7 days prior to registration
* Ability to understand and willingness to sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent document prior to registration
* Willingness and ability of subject to comply to study requirements

Exclusion Criteria:

* Patients may not be receiving any other investigational agents; a 2 week washout period for investigational agents is required before registration
* Patients with clinically symptomatic brain metastases or who required treatment for brain metastases within 4 weeks of registration (stable sequelae acceptable if treatment has been completed; these lesions cannot be used as target lesions)
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to denosumab are not eligible (i.e. same class of drugs) (Note: prior bisphosphonates are allowed; patients could have received bisphosphonates or be bisphosphonate-naive; patients who were previously on bisphosphonates can be enrolled in the study, as long as they have a wash-out period of 2 weeks prior to registration)
* Patients who are on corticosteroids or immunosuppressant's are not eligible; a 2 week wash-out period for is required before registration
* Patients who have a known additional malignancy that is progressing or requires active treatment are not eligible; patients who have had a prior diagnosis of cancer and if it has been < 3 years since their last treatment are also not eligible; NOTE: exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension (defined as 160/90 mmHg for 3 consecutive readings 2-5 mins apart) that is not controlled on medication
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Subject is pregnant or breast feeding, or planning to become pregnant within 5 months after the end of treatment
* Known human immunodeficiency virus (HIV)-positive patients who are on combination antiretroviral therapy; (this is because of the potential for pharmacokinetic interactions with denosumab)
* No known prior history or current evidence of osteonecrosis/osteomyelitis of the jaw
* No known prior history or current evidence of untreated local gum or oral infection
* No known/planned active dental or jaw condition which requires oral surgery, including tooth extraction
* No known non-healed dental/oral surgery, including tooth extraction
* Patients have planned invasive dental procedures during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarika Jain, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Northwestern University- Lake Forest Hospital, Lake Forest, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for enrollment on March 23, 2017 with an accrual goal of 42 patients. The first patient started treatment on study October 19, 2017. The study closed permanently to enrollment on March 6 2018 with one patient enrolled, due to low accrual and before total accrual to the study could be met.
Period: 3 Cycles of Treatment
Arm/Group | Treatment (Denosumab)
Started | 1
Completed | 1
Not Completed | 0
Period: Follow up for 2 Years
Arm/Group | Treatment (Denosumab)
Started (Everyone that receives treatment on study goes into the follow up phase) | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Denosumab)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Patients With Reduction in CTCs
Description: Assess the effect of denosumab in Her2/neu negative ER+ and/ or PR+ metastatic breast cancer patients who are in Partial Response (PR) or Stable Disease (SD) after starting systemic therapy with bone metastases and ≥ 5 CTCs by measuring the fraction of patients with reduction in CTCs.
Time Frame: Up to 3 months
Population: Data was not collected or analyzed for this outcome measure. The study was terminated early with only 1 patient enrolled.
Arm/Group | Treatment (Denosumab)
Number analyzed (Participants) | 0

2. Secondary Outcome: Percent Change in CTCs
Description: Evaluate the effect of denosumab on CTCs enumeration by assessing the percent change from baseline.
Time Frame: Baseline up to 3 months
Population: as for outcome 1
Arm/Group | Treatment (Denosumab)
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Progression Free Survival
Description: Assess median progression free survival (m-PFS) using statistical analysis evaluating the relationship between longitudinal CTC counts and PFS. PRS will be measured from the time of treatment up until progressive disease.
Time Frame: Up to 2 years
Population: as for outcome 1
Arm/Group | Treatment (Denosumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 3 cycles of treatment and up to 30 days past the last treatment, where 1 cycle of treatment equals 28 days.
Arm/Group | Treatment (Denosumab)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Denosumab) (N=1)
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hoarsness (Respiratory, thoracic and mediastinal disorders) | 1
Hypoabuminemia (Metabolism and nutrition disorders) | 1
Alkaline phosphatase increased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early with only 1 patient enrolled due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT03070002/Prot_SAP_000.pdf